CLINICAL TRIAL: NCT03623529
Title: A Randomised, Placebo-controlled, Double-Blind, Multicentre Efficacy and Safety Study of LJPC-501 in Paediatric Patients > 2 to 17 Years of Age With Catecholamine-Resistant Hypotension Associated With Distributive Shock
Brief Title: A Study of LJPC-501 in Paediatric Patients With Hypotension Associated With Distributive or Vasodilatory Shock
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LJ501-CRH04
Record Dates: First submitted 2018-06-29; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Catecholamine-resistant Hypotension (CRH); Distributive Shock; High Output Shock; Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Angiotensin I; Angiotensin II; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Comparator: LJPC-501 (Experimental): LJPC-501 Angiotensin II Solution for infusion
  Interventions: Drug: LJPC-501 (angiotensin II)
- Placebo Comparator: Placebo (Placebo Comparator): 0.9% sodium chloride solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LJPC-501 (angiotensin II) — Angiotensin II is a peptide hormone naturally produced by the body that regulates blood pressure via vasoconstriction and sodium reabsorption.
  Arms: Active Comparator: LJPC-501
Drug: Placebo — Placebo Arm
  Other Names: 0.9% sodium chloride solution
  Arms: Placebo Comparator: Placebo

SUMMARY:
The objective of this study is to evaluate the effect of LJPC-501 infusion on mean arterial pressure (MAP) as assessed by standard of care vasopressor dose reduction in pediatric patients with catecholamine-resistant hypotension (CRH). In addition, this study will evaluate the safety and tolerability of LJPC-501 in pediatric patients, evaluate changes in catecholamine and other vasopressor doses over time, evaluate the change in MAP over time, and the change in Pediatric Logistic Organ Dysfunction-2 (PELOD-2) scores.

ELIGIBILITY:
Inclusion Criteria:

Male and female paediatric patients with catecholamine-resistant hypotension associated with distributive shock.

1. Paediatric patients > 2 years (ie, > 24 months) to < 18 years of age at enrolment.
2. Patients requiring a sum norepinephrine-equivalent dose > 0.1 μg/kg/min to maintain age-appropriate target MAP for a minimum of 2 hours and a maximum of 48 hours prior to initiation of study drug.
3. Patients must have a clinical diagnosis of distributive shock in the opinion of the treating team and the Investigator.
4. Patients are required to have central venous access, which is expected to remain present for the duration of study drug treatment.
5. Patients are required to have an indwelling arterial line, which is expected to remain present for at least the first 48 hours of study drug treatment.
6. Patients must have received at least 40 mL/kg of crystalloid or colloid equivalent over the initial 24-hour resuscitation period, and must be adequately volume resuscitated in the opinion of the Investigator, prior to starting study drug.
7. Parent(s) or legal guardian(s) is willing and able to provide informed consent and assist the patient in complying with all protocol requirements.

Exclusion Criteria:

1. Patients who are ≤ 2 years (24 months) of age or ≥ 18 years of age at enrolment.
2. Patients with a standing Do Not Resuscitate order.
3. Patients diagnosed with acute occlusive coronary syndrome requiring pending intervention.
4. Patients on veno-arterial (VA) extracorporeal membrane oxygenation (ECMO).
5. Patients who have been on veno-venous (VV) ECMO for less than 6 hours.
6. Patients with a clinical suspicion of cardiogenic shock based on echocardiogram.
7. Patients who have a history of asthma or are currently experiencing bronchospasm requiring the use of inhaled bronchodilators and who are not mechanically ventilated.
8. Patients with acute mesenteric ischaemia or a history of mesenteric ischaemia.
9. Patients with active bleeding AND an anticipated need of multiple transfusions (within 48 hours of Screening).
10. Patients with active bleeding AND haemoglobin < 7 g/dL.
11. Patients with an expected lifespan of < 12 hours or expected withdrawal of life support within 24 hours of Screening.
12. Patients with a known allergy to mannitol.
13. Patients who are currently participating in another clinical trial using an investigational drug not approved in that member country unless specifically approved by the Sponsor.
14. Patients of childbearing potential who are known to be pregnant at the time of Screening.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who have a >/= 50% reduction in norepinephrine equivalent doses (NED) | Hour 3

SECONDARY OUTCOMES:
Effect on Paediatric Logistic Organ Dysfunction-2 (PELOD-2) based on treatment with LJPC-501 | Baseline, Hour 24 and Hour 48
  Change in PELOD-2 score from baseline to 24 hours and 48 hours after start of LJPC-501. The PELOD-2 score is the sum of 5 individual item scores that totals 0-31 points. A higher PELOD-2 score represents a worse outcome.
Effect on total catecholamine doses administered based on treatment with LJPC-501 | Baseline, Hour 24 and Hour 48
  Change in total catecholamine doses administered from baseline to 24 hours and 48 hours after start of LJPC-501.
Effect on mean arterial pressure (MAP) based on treatment with LJPC-501 | Baseline, Hour 3, Hour 24, and Hour 48
  Change in MAP from baseline to 3 hours, 24 hours and 48 hours after start of LJPC-501
Effect on heart rate based on treatment with LJPC-501 | Baseline to Hour 3, Hour 24, and Hour 48
  Change in heart rate from baseline to 3 hours, 24 hours and 48 hours after start of LJPC-501
Assessment of safety based on number of patients with treatment emergent adverse events based on treatment with LJPC-501 | Day 7
Assessment of tolerability based on the effect on clinical chemistry parameters based on treatment with LJPC-501 | Hour 24 and Hour 48
  Safety data for clinical chemistry parameters including ALT, AST, ALP, total bilirubin, direct bilirubin, creatinine, BUN, lactate, phosphorous, glucose, albumin, calcium, bicarbonate, chloride, sodium, potassium, magnesium

CONTACTS AND LOCATIONS:
Locations (2):
- Investigational Site, Brussels, Belgium
- Investigational Site, Vilnius, Lithuania